CLINICAL TRIAL: NCT01491347
Title: Brain Derived Neurotrophic Factor Serum Levels Evolution During the Six Months Following After Alcohol Withdrawal in Alcohol-dependent Subjects in Relation to Abstinence
Brief Title: Brain Derived Neurotrophic Factor Serum Levels Evolution During the Six Months After Alcohol Withdrawal
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Esquirol (Other)
Responsible Party: Principal Investigator, Philippe Nubukpo, MD, PhD, Centre Hospitalier Esquirol
Other Study IDs: 2011-A00452-39
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Alcohol Dependence
Keywords: BDNF; withdrawal; alcohol; psychiatry
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- alcohol dependent

SUMMARY:
Alcohol dependence is accompanied by several neurological mechanisms involving neuronal plasticity and neoneurogenesis, requiring Brain Derived Neurotrophic factor (BDNF) synthesis.

The investigators found that serum BDNF levels in alcohol-dependent subjects increased to a greater extent in subjects who had remained abstinent at 6 months after withdrawal than in subjects who had relapse.

To verify if the BDNF serum levels variation is linked to the way that abstinence is installed, wthe investigators will measure BDNF serum levels in alcohol dependent subjects at the moment of withdrawal, and 14, 28 days, and 2, 4, and 6 months after to establish its evolution in relation to alcohol consumption, and other clinical characteristics : depression intensity, anxiety, alcohol craving, biological markers of alcohol consumption or toxicity. Monitoring serum BDNF concentrations in link with other clinical data could help to characterize alcohol dependence profiles in clinical practice, help predict relapses, and assist in adjusting care to prevent difficulties in alcohol withdrawal.

DETAILED DESCRIPTION:
A total of 205 patients will be recruited at their hospitalization time for alcohol withdrawal during a 18 months period. The follow-up at 14, 28 days, 2, 4, 6 months after alcohol withdrawal will assess their BDNF serum levels, the levels of carbohydrate deficient transferrin (CDT), gamma glutamyl transferase (GGT), urinary ethylglucuronide (EtG), and the scores to the Beck Depression Inventory (BDI), the Montgomery Asberg depression scale (MADRS), the Hamilton'anxiety scale (HAM-A), the Obsessive Compulsive Drinking Scale (OCDS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of alcohol dependence according to the DSM-IV-TR
* Request for withdrawal

Exclusion Criteria:

* Age < 18 years
* Psychiatric co-morbidity in an evoluting stage and predominant on the addiction trouble
* Characterized (diagnosed) neurological co-morbidity
* Severe somatic pathology and / or with fatal predicted outcome in the year (cancer...)
* Inability to answer the questionnaires
* pregnancy
* neuroleptic or antidepressant treatment established for less than 3 months
* anti-retroviral treatment
* absence of consent, judiciary protection, hospitalization under constraint, - absence of health insurance.
* Residence at more than 80 km from the study center
* Participation to an other biomedical study during the 6 months of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with alcohol dependance diagnosis according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR), and asking for alcohol withdrawal in hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 389 (Actual)
Dates: Start 2011-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
BDNF serum levels variations between alcohol withdrawal and 14-, 28- days, 2-, 4- and 6- months after in relation to abstinence at 6 months. | 6 months

SECONDARY OUTCOMES:
Search of a correlation between serum BDNF levels and alcohol consumption marker (CDT), GGT, EtG at 28 days 2, 4, and 6 months after alcohol withdrawal. | 6 months
Search of a correlation between serum BDNF levels and the scores to psychometric scales : BDI, MADRS, HAM-A, OCDS, at 28 days 2, 4, and 6 months after alcohol withdrawal. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Nubukpo, MD, PhD, Principal Investigator — Centre Hospitalier Esquirol
Locations (4):
- France (4):
  - Clinique Saint Maurice, La Jonchère
  - Centre Hospitalier Esquirol, Limoges
  - Centre Hospitalier de Vauclaire, Montpon-Ménestérol
  - Centre Hospitalier La Vallette, Saint-Vaury

REFERENCES:
- [Background] Costa MA, Girard M, Dalmay F, Malauzat D. Brain-derived neurotrophic factor serum levels in alcohol-dependent subjects 6 months after alcohol withdrawal. Alcohol Clin Exp Res. 2011 Nov;35(11):1966-73. doi: 10.1111/j.1530-0277.2011.01548.x. Epub 2011 Aug 16. PMID 21848960
- [Derived] Pareaud M, Girard M, Nubukpo P. Factors for Maintaining Abstinence at 2 and 6 Months After Alcohol Withdrawal. J Psychiatr Pract. 2021 Jan 21;27(1):2-13. doi: 10.1097/PRA.0000000000000522. PMID 33438862